CLINICAL TRIAL: NCT02441569
Title: Common Engagement Strategies (Common Factors) for Childhood Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P20MH086048 (NIH)
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Common factors intervention (Experimental): Children and parents in this arm will be cared for by a provider who has received brief training in common factors patient engagement skills (the intervention) for use in addition to standard anxiety-related advice. Thus this arm will receive common factors engagement training for provider.
  Interventions: Behavioral: Common factors engagement training for provider; Behavioral: Standard pediatric advice for childhood anxiety
- Control (Active Comparator): Children and parents in this arm will be cared for by a provider who is able to offer standard pediatric anxiety-related advice (the control intervention). Families will receive standard pediatric advice for childhood anxiety.
  Interventions: Behavioral: Standard pediatric advice for childhood anxiety

INTERVENTIONS:
Behavioral: Common factors engagement training for provider — Primary care providers have received brief training in communication skills designed to promote family engagement in care including understanding of treatment and empowerment.
  Arms: Common factors intervention
Behavioral: Standard pediatric advice for childhood anxiety — Providers will be free to use their existing knowledge of anxiety problems to offer routine counseling.

SUMMARY:
This trial examines the effectiveness of training pediatric primary care providers (nurse practitioners, doctors) to use of strategies that enhance family/youth empowerment and engagement during office visits for children with mild to moderate problems with anxiety. Children coming for routine care at one clinic are screened for anxiety symptoms and seen by either a specially trained provider or one of the clinic's other regular staff members.

DETAILED DESCRIPTION:
Children who are thought to have mild to moderate anxiety will, via their parents, be offered the opportunity to receive treatment from their pediatric primary care provider. Providers will either use their existing anxiety approaches or will use those approaches combined with extra communication skills designed to promote patient and parent engagement in care. Children will be seen for up to 4 30-minute visits at 2 week intervals, with a follow-up telephone call 3 months later to asses the impact of treatment. Children with more severe anxiety (or those whose parents so desire) will be referred for specialized mental health care.

ELIGIBILITY:
Inclusion Criteria:

* Coming for well-child visit to designated clinical site;
* SCARED score 25 or greater

Exclusion Criteria:

* acute medical illness, SCARED 40 or greater

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The Screen for Child Anxiety Related Emotional Disorders (SCARED) | 3 months
  Re-test on short inventory of anxiety-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Wissow, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Georgetown University Pediatric Clinic, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No